CLINICAL TRIAL: NCT03394625
Title: Evaluation of Marginal Bone Loss in Immediate Implant Placement in Maxillary Esthetic Zone Using Socket Shield Technique Versus Xenogenous Bone Substitute Material
Brief Title: Evaluate Marginal B. Loss in Immediate Implant Placement in Maxillary Esthetic Zone Using Socket Shield Versus Xenograft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Ibrahim Shaalan, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Shaalancuimplant
Record Dates: First submitted 2017-12-27; First posted 2018-01-09 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Marginal Bone Loss in Socket Shield Technique
Keywords: Socket Shield; immediate implant; ridge preservation
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate implant placement using socket shield technique (Experimental): Socket shield technique is a recent technique which is by sectioning the root and extraction of palatal part and leaving buccal part of the root with its attachment of periodontal ligament and vascularization still intact then placing implant in palatal socket.
  Interventions: Procedure: Socket shield technique
- immediate implant placement using xenograft material (Active Comparator): placing xenograft material in gap between implant and buccal bone
  Interventions: Procedure: using Xenograft material

INTERVENTIONS:
Procedure: Socket shield technique — Socket shield technique is a recent technique which is by sectioning the root and extraction of palatal part and leaving buccal part of the root with its attachment of periodontal ligament and vascularization still intact then placing implant in palatal socket.
  Arms: immediate implant placement using socket shield technique
Procedure: using Xenograft material — placing xenograft material in gap between the implant and the buccal plate of bone
  Arms: immediate implant placement using xenograft material

SUMMARY:
Anterior maxilla (Esthetic zone) is very challenging area because of thin buccal plate of bone. After tooth extraction physiological process occur causing alteration of bone and soft tissue so, delayed placement of implant lead to loss of bone height and width. Immediate placement of implant is become essential to preserve the bone and soft tissue from loss.

Socket shield technique is a recent technique which is by sectioning the root and extraction of palatal part and leaving buccal part of the root with its attachment of periodontal ligament and vascularization still intact then placing implant in palatal socket. This technique allow preservation of buccal plate of bone and soft tissue with minimum loss allowing better result in esthetic zone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with badly broken teeth in upper esthetic zone with intact periodontal condition indicated for extraction, presence of at least 4 mm of bone beyond the root apex to guarantee implant primary stability, implant placement within the alveoli confines.
* Both sexes.
* No intraoral soft and hard tissue pathology.
* Physically able to tolerate conventional surgical and restorative procedures.
* Signing of an informed consent form.

Exclusion Criteria:

* Presence of fenestrations or dehiscence of the residual bony walls after extraction.
* Heavy smokers more than 20 cigarettes per day .(24)
* Patients with systemic disease that may affect normal healing e.g. uncontrolled diabetes.
* Psychiatric problems e.g. severe bruxism.
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site.
* Active infection in the teeth to be treated
* Vertical root fractures with displacement in the teeth of the surgical area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-12-20 (Estimated)

PRIMARY OUTCOMES:
marginal bone loss | 4 months
  will be measured from CBCT using Blue-sky software built-in linear measuring tool by millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt